CLINICAL TRIAL: NCT00569933
Title: Audio Recording for Improved Surgical Outcome
Brief Title: Audio Recording for Improved Surgical Outcome (ARISO)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, James H. Stewart, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 06-002226
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Osteoarthritis
Keywords: Hip Surgery; Perioperative; suggestions/imagery
MeSH Terms: conditions — Osteoarthritis | interventions — Sound Recordings

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A/B/C (Other): Patients are randomized to voice/music/ or no CD
  Interventions: Behavioral: Audio recording

INTERVENTIONS:
Behavioral: Audio recording — Using audio recording to investigate if possitive affirmations help with pain management and other post of compllication.

SUMMARY:
Use of audio recordings (with suggestions and imagery for a better surgical outcome) studied in orthopedic patients.

DETAILED DESCRIPTION:
Pt undergoing orthopedic surgery are randomized into 3 groups. These interventionals will be listening to CD recording just prior to and during orthopedic surgery. The 2nd group will be listening to a recording before and during surgery without any positive suggestions. The 3rd group will be receiving usual care. Prior to hospital discharge patients will fill out a questionaire assessing their perception of their surgery and hospital stay. Pt. charts will be reviewed for use of pain, sleep, anesthesia and nausea medication and for the number of units of blood transfused. Pt. outcomes will be asssessed with this data.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total hip replacement under reginal anethesia at Mayo Clinic in Jacksonville, Fl.
* Willingness to sign consent.
* Age 18 or greater.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Post Op pain | Day 1 to 3

SECONDARY OUTCOMES:
Blood Loss, Nausea, sleep | Day 1 to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: James H. Stewart, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States